CLINICAL TRIAL: NCT00164177
Title: A Preliminary Evaluation Of The Efficacy Of HalfLYTELY® For Bowel Cleansing Before Virtual Colonoscopy (VC) and Conventional Colonoscopy (CC).
Brief Title: Evaluation Of The Efficacy Of HalfLYTELY For Bowel Cleansing Before Virtual Colonoscopy and Conventional Colonoscopy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: F38-VC-002
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy
Keywords: virtual colonoscopy; colonoscopy preparation; bowel prep

INTERVENTIONS:
Drug: HalfLytely

SUMMARY:
To evaluate the efficacy of standard HalfLYTELY® as a bowel cleansing preparation for adult patients undergoing virtual colonoscopy (VC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for routinely accepted indications, Evaluation of BE results, GI bleeding, Anemia of unknown etiology, Neoplastic disease surveillance, Endosonography, Inflammatory bowel disease (except as noted below), Unknown diarrhea etiology, Prior Polypectomy, Laser therapy, Foreign body removal and decompression (except as noted below).
* 18 years of age or older.
* Otherwise in good health, as determined by physical exam and medical history.
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, or vasectomized spouse)
* Subject has read and signed the written informed consent document prior to study participation

Exclusion Criteria:

* Subjects with known or suspected bowel perforation or obstruction, inflammatory bowel disease, ileus, acute alimentary tract surgery, significant gastroparesis or gastric outlet obstruction, appendicitis, gastric retention, toxic colitis, toxic megacolon or rectal bleeding.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects with uncontrolled cardiovascular disease
* Subjects who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational clinical surgical, drug or device study within the past 30 days.
* Subjects who are pregnant or lactating.
* Subjects who are allergic to Polyethyleneglycol.
* Subjects receiving non-study laxatives, antacids and prokinetic agents during the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-10; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of the preparation to produce a degree of fecal matter and residual liquid that would not interfere with VC or CC.

SECONDARY OUTCOMES:
Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: H. Paul Hatten, Jr., MD, Principal Investigator — Indian River Radiology
Locations (1):
- Vero Beach, Florida, United States